CLINICAL TRIAL: NCT03070392
Title: A Phase II Randomized, Open-label, Multi-center Study of the Safety and Efficacy of IMCgp100 Compared With Investigator Choice in HLA-A*0201 Positive Patients With Previously Untreated Advanced Uveal Melanoma
Brief Title: Safety and Efficacy of IMCgp100 Versus Investigator Choice in Advanced Uveal Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Immunocore Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMCgp100-202
Expanded Access: NCT04960891 (Available)
Record Dates: First submitted 2017-02-14; First posted 2017-03-03 (Actual); Results first posted 2021-09-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Uveal Melanoma
Keywords: Melanoma; Uveal Cancer; IMCgp100; Immunotherapy; Tebentafusp; Ocular Melanoma; Eye Melanoma; Uveal Melanoma; Gp100; TCR; Dacarbazine; Ipilimumab; Pembrolizumab; Bispecific T cell receptor fusion protein; ImmTAC; Immune mobilizing monoclonal T cell receptor against cancer; Kimmtrak
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Dacarbazine; Ipilimumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMCgp100 (tebentafusp, Kimmtrak) (Experimental): Biologic:IMCgp100 (Soluble gp 100-specific T cell receptor with anti - CD3 scFV: IMCgp100)
  Interventions: Biological: IMCgp100
- Investigator's Choice (Active Comparator): 1 of 3 Investigator's Choice options: Systemic Dacarbazine
  1 of 3 Investigator's Choice options: Systemic Ipilimumab
  1 of 3 Investigator's Choice options: Systemic Pembrolizumab
  Interventions: Drug: Dacarbazine; Biological: Ipilimumab; Biological: Pembrolizumab

INTERVENTIONS:
Biological: IMCgp100 — IMCgp100 is to be administered at 20 mcg cycle 1 day1, then 30 mcg cycle 1 day 8, then 68 mcg cycle 1 day 15 and weekly thereafter by IV infusion over 15 minutes until confirmed disease progression or unacceptable toxicity
  Arms: IMCgp100 (tebentafusp, Kimmtrak)
Drug: Dacarbazine — Dacarbazine is to be administered at 1,000 mg/m2 of body surface area IV infusion every 3 weeks until disease progression or unacceptable toxicity
  Other Names: DTIC-Dome; DTIC; DIC; Imidazole Carboxamide
  Arms: Investigator's Choice
Biological: Ipilimumab — Ipilimumab is to be administered at 3 mg/kg IV infusion over 90 minutes every 3 weeks for a total of 4 treatments
  Other Names: Yervoy
  Arms: Investigator's Choice
Biological: Pembrolizumab — Pembrolizumab is to be administered at 2 mg/kg IV infusion up to a maximum of 200 mg administered Intravenously over 30 minutes every 3 weeks or 200 mg fixed dose administered intravenously every 3 weeks where approved locally until confirmed disease progression or unacceptable toxicity
  Other Names: Keytruda
  Arms: Investigator's Choice

SUMMARY:
To evaluate the overall survival of HLA-A*0201 positive adult patients with previously untreated advanced UM receiving IMCgp100 compared to Investigator's Choice of dacarbazine, ipilimumab, or pembrolizumab.

DETAILED DESCRIPTION:
This Phase II study is designed to evaluate the safety and efficacy of IMCgp100 compared with Investigator's Choice (dacarbazine, ipilimumab or pembrolizumab) in HLA-A*0201 positive adult patients with advanced UM treated in the first line setting with no prior systemic or liver-directed chemo-, radio- or immune-therapy administered in the advanced setting (prior surgical resection of liver metastases and adjuvant systemic therapy are acceptable). Comparison of the IMCgp100 efficacy results in this Phase II study will be made with the concurrently randomized arm (Investigator's Choice) with a primary endpoint of overall survival (OS) and secondary efficacy endpoints of progression-free survival (PFS), objective response rate (ORR), duration of response (DOR), and disease control rate (DCR).

ELIGIBILITY:
Inclusion Criteria

1. Male or female participants age ≥ 18 years of age at the time of informed consent
2. Ability to provide and understand written informed consent prior to any study procedures
3. Histologically or cytologically confirmed metastatic UM
4. Must meet the following criteria related to prior treatment:

   * No prior systemic therapy in the metastatic or advanced setting including chemotherapy, immunotherapy, or targeted therapy
   * No prior regional, liver-directed therapy including chemotherapy, radiotherapy, or embolization
   * Prior surgical resection of oligometastatic disease is allowed
   * Prior neoadjuvant or adjuvant therapy is allowed provided administered in the curative setting in participants with localized disease. Participants may not be re-treated with an Investigator's Choice therapy that was administered as adjuvant or neoadjuvant treatment. Additionally, participants who have received nivolumab as prior adjuvant/neoadjuvant treatment should not receive pembrolizumab as Investigator's Choice therapy.
5. HLA A*0201 positive by central assay
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 at Screening
7. Participants have measurable disease or non-measurable disease according to RECIST v1.1
8. All other relevant medical conditions must be well-managed and stable, in the opinion of the investigator, for at least 28 days prior to first administration of study drug

Exclusion Criteria

1. Out-of-range laboratory values
2. History of severe hypersensitivity reactions (eg, anaphylaxis) to other biologic drugs or monoclonal antibodies
3. Clinically significant cardiac disease or impaired cardiac function,
4. Presence of symptomatic or untreated central nervous system (CNS) metastases, or CNS metastases that require doses of corticosteroids within the prior 3 weeks to study Day 1. Participants with brain metastases are eligible if lesions have been treated with localized therapy and there is no evidence of PD for at least 4 weeks by magnetic resonance imaging (MRI) prior to the first dose of study drug
5. Active infection requiring systemic antibiotic therapy. Participants requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to the first dose of study drug
6. Known history of human immunodeficiency virus infection (HIV). Testing for HIV status is not necessary unless clinically indicated
7. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection per institutional protocol. Testing for HBV or HCV status is not necessary unless clinically indicated or the patient has a history of HBV or HCV infection
8. Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to study treatment; completely resected basal cell and squamous cell skin cancers; any malignancy considered to be indolent and that has never required therapy; and completely resected carcinoma in situ of any type
9. Any medical condition that would, in the investigator's or Sponsor's judgment, prevent the participants participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results
10. Participants receiving systemic steroid therapy or any other systemic immunosuppressive medication at any dose level, as these may interfere with the mechanism of action of study treatment. Local steroid therapies (eg, otic, ophthalmic, intra-articular, or inhaled medications) are acceptable
11. History of adrenal insufficiency
12. History of interstitial lung disease
13. History of pneumonitis that required corticosteroid treatment or current pneumonitis
14. History of colitis or inflammatory bowel disease
15. Major surgery within 2 weeks of the first dose of study drug (minimally invasive procedures such as bronchoscopy, tumor biopsy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery and are not exclusionary)
16. Radiotherapy within 2 weeks of the first dose of study drug, with the exception of palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass
17. Use of hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF, M-CSF) ≤ 2 weeks prior to start of study drug. An erythroid-stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment and the patient is not red blood cell transfusion dependent
18. Pregnant, likely to become pregnant, or lactating women (where pregnancy is defined as the state of a female after conception and until the termination of gestation)
19. Women of childbearing potential who are sexually active with a non-sterilized male partner, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception during study treatment (defined in Section 6.7), and must agree to continue using such precautions for 6 months after the final dose of investigational product; cessation of birth control after this point should be discussed with a responsible physician. Highly effective methods of contraception are described in Section 6.7
20. Male participants must be surgically sterile or use double barrier contraception methods from enrollment through treatment and for 6 months following administration of the last dose of study drug
21. Participant who are in an institution due to official or judicial order.
22. Participant who are the investigator or any subinvestigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in the conduct of the study.
23. Contraindication for treatment with Investigator's Choice alternatives (dacarbazine, ipilimumab and pembrolizumab) as per applicable labelling. Participant may have a contraindication to 1 or 2 of the choices if he/she is a candidate for dosing with at least 1 Investigator's Choice and meets all other study eligibility criteria.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Immunocore Medical Information, Study Director — Immunocore Ltd
Locations (57):
- United States (23):
  - UCLA Medical Center, Los Angeles, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Byers Eye Institute, Stanford University, Palo Alto, California
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Health System, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Portland Providence Medical Center, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Houston Methodist Cancer Center, Houston, Texas
- Australia (3):
  - Saint Vincents Hospital, Darlinghurst, New South Wales
  - Central Adelaide Local Health Network, Royal Adelaide Hospital Cancer Center, Adelaide, South Australia
  - Peter MacCallum Cancer Center, Melbourne, Victoria
- Belgium (2):
  - Institut Roi Albert II Cliniques Universitaires St-Luc, Brussels
  - Universite Catholique de Louvain Centre du Cancer, Medical Oncology, Brussels
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto
- France (2):
  - Centre Atoine Lacassagne, Nice
  - Institut Curie, Paris
- Germany (7):
  - Universitaetsklinikum Koeln Dermatologie und Venerologie, Cologne, North Rhine-Westphalia
  - Charite - Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - University Hospital Essen, Essen
  - University of Hamburg, Hamburg
  - Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Klinik und Poliklinik für Dermatologie und Allergologie, Munich
- Italy (2):
  - Fondazione ICCRS, Milan
  - Istituto Nazionale Tumori - IRCCS Fondazione "G. Pascale" - UOC Melanoma, Immunoterapia Oncologica e Terapie Innovative, Napoli
- LUMC Medical Oncology, Leiden, Netherlands
- Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw, Poland
- Russia (2):
  - Federal State Budgetary Institution N.N. Blokhin National Medical Research Center of Oncology, Moscow
  - Federal State Budget Institution National Medical Research Center of Oncology, Saint Petersburg
- Spain (5):
  - Institut Catala d'Oncologia (ICO) - L'Hospitalet, L'Hospitalet de Llobregat, ES-Spain
  - Hospital Universitario La Paz, Madrid, ES-Spain
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, ES-Spain
  - Hospital Universitario General de Valencia, Valencia, ES-Spain
  - Hospital Universitario Virgen Macarena, Seville
- University of Zurich Hospital, Zurich, Switzerland
- Ukraine (3):
  - Dnipropetrovsk State Medical Academy, Dnipro
  - Kyiv Munitipal Hospital, Kyiv
  - Uzhhorod Central City Clinical Hospital, Uzhhorod
- United Kingdom (3):
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - The Clatterbridge Cancer Centre, Bebington, Wirral
  - Beatson West of Scotland Cancer Centre, Glasgow

REFERENCES:
- [Derived] Hassel JC, Piperno-Neumann S, Rutkowski P, Baurain JF, Schlaak M, Butler MO, Sullivan RJ, Dummer R, Kirkwood JM, Orloff M, Sacco JJ, Ochsenreither S, Joshua AM, Gastaud L, Curti B, Piulats JM, Salama AKS, Shoushtari AN, Demidov L, Milhem M, Chmielowski B, Kim KB, Carvajal RD, Hamid O, Collins L, Ranade K, Holland C, Pfeiffer C, Nathan P. Three-Year Overall Survival with Tebentafusp in Metastatic Uveal Melanoma. N Engl J Med. 2023 Dec 14;389(24):2256-2266. doi: 10.1056/NEJMoa2304753. Epub 2023 Oct 21. PMID 37870955
- [Derived] Nathan P, Hassel JC, Rutkowski P, Baurain JF, Butler MO, Schlaak M, Sullivan RJ, Ochsenreither S, Dummer R, Kirkwood JM, Joshua AM, Sacco JJ, Shoushtari AN, Orloff M, Piulats JM, Milhem M, Salama AKS, Curti B, Demidov L, Gastaud L, Mauch C, Yushak M, Carvajal RD, Hamid O, Abdullah SE, Holland C, Goodall H, Piperno-Neumann S; IMCgp100-202 Investigators. Overall Survival Benefit with Tebentafusp in Metastatic Uveal Melanoma. N Engl J Med. 2021 Sep 23;385(13):1196-1206. doi: 10.1056/NEJMoa2103485. PMID 34551229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 378 patients were randomly assigned (2:1) to Tebentafusp (n=252) or Investigator's Choice (n=126) at 58 sites in 14 countries.
Pre-assignment Details: The data cut-off date for this analysis was 13 October 2020. Combining participants into a single group as part of the Investigator's Choice arm was pre-specified as part of the study design.
Groups:
- Tebentafusp: Tebentafusp administered at 20 mcg at Cycle 1 Day 1, 30 mcg at Cycle 1 Day 8, and 68 mcg at Cycle 1 Day 15 by IV infusion and weekly thereafter.
- Investigator's Choice: Dacarbazine: Dacarbazine administered at 1,000 mg/m^2 of body surface area IV infusion every 3 weeks until confirmed disease progression or unacceptable toxicity.
- Investigator's Choice: Ipilimumab: Ipilimumab administered at 3 mg/kg IV infusion over 90 minutes every 3 weeks for a total of 4 treatments.
- Investigator's Choice: Pembrolizumab: Pembrolizumab administered at 2 mg/kg IV infusion over 30 minutes every 3 weeks or 200 mg fixed dose administered intravenously every 3 weeks where approved locally until confirmed disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Tebentafusp | Investigator's Choice: Dacarbazine | Investigator's Choice: Ipilimumab | Investigator's Choice: Pembrolizumab
Started | 252 | 7 | 16 | 103
Completed | 0 | 0 | 10 | 0
Not Completed | 252 | 7 | 6 | 103
Not completed — Not Treated | 7 | 0 | 3 | 12
Not completed — Death | 3 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 3
Not completed — Physician Decision | 1 | 0 | 0 | 2
Not completed — Progressive Disease | 154 | 6 | 2 | 70
Not completed — Adverse Event | 6 | 1 | 1 | 3
Not completed — Alternate anticancer treatment | 1 | 0 | 0 | 1
Not completed — Ongoing | 73 | 0 | 0 | 11

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) Analysis Set comprises all participants assigned to treatment analyzed by the treatment assignment whether or not the participant received the assigned treatment. Combining participants into a single group as part of the Investigator's Choice arm was pre-specified as part of the study design.
Groups:
- Investigator's Choice: 1 of 3 Investigator's Choice options: Systemic Dacarbazine, Ipilimumab or Pembrolizumab. Dacarbazine: administered at 1,000 mg/m2 of body surface area IV infusion every 3 weeks until disease progression or unacceptable toxicity; Ipilimumab: administered at 3 mg/kg IV infusion over 90 minutes every 3 weeks for a total of 4 treatments; Pembrolizumab: administered at 2 mg/kg IV infusion up to a maximum of 200 mg administered Intravenously over 30 minutes every 3 weeks or 200 mg fixed dose administered intravenously every 3 weeks where approved locally until confirmed disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Tebentafusp | Investigator's Choice | Total
Number analyzed (Participants) | 252 | 126 | 378
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (11.9) | 63.6 (10.7) | 62.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 64 | 188
  Male | 128 | 62 | 190
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 222 | 107 | 329
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 30 | 18 | 48

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Overall Survival
Description: Overall survival is defined as the time from randomization to date of death due to any cause.
Time Frame: From randomization to the data cut off date of 13-Oct-2020; median follow-up duration was 14.1 months.
Population: The Intent-to-treat (ITT) Analysis Set comprises all participants assigned to treatment analyzed by the treatment assignment whether or not the participant received the assigned treatment. Combining participants into a single group as part of the Investigator's Choice arm was pre-specified as part of the study design; therefore, data per different treatments were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tebentafusp | Investigator's Choice
Number analyzed (Participants) | 252 | 126
Months | 21.7 [18.6 to 28.6] | 16.0 [9.7 to 18.4]
Statistical Analysis 1: Comparison: Tebentafusp vs Investigator's Choice; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.37 to 0.71]

2. Secondary Outcome: Safety: Number of Participants With Treatment Emergent Adverse Events
Description: Safety was defined as the number of participants with treatment emergent adverse events, including laboratory abnormalities, ECG changes, and/or physical examination findings.
Time Frame: Safety was assessed from informed consent through 90 days after end of treatment, up to 36 months.
Population: The Safety Analysis Set includes all randomized participants who received at least 1 full or partial dose of tebentafusp or investigator's choice. Combining participants into a single group as part of the Investigator's Choice arm was pre-specified as part of the study design; therefore, data per different treatments were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Tebentafusp | Investigator's Choice
Number analyzed (Participants) | 245 | 111
Participants | 245 | 105

3. Secondary Outcome: Efficacy: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from randomization to the date of progression (RECIST v1.1) or death due to any cause.
Time Frame: PFS was assessed every 3 months from randomization until disease progression or death, up to 36 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tebentafusp | Investigator's Choice
Number analyzed (Participants) | 252 | 126
Months | 3.3 [3.0 to 5.0] | 2.9 [2.8 to 3.0]
Statistical Analysis 1: Comparison: Tebentafusp vs Investigator's Choice; Test type: Superiority; p = 0.0139, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.58 to 0.94]

4. Secondary Outcome: Quality-of-Life: Change From Baseline in EQ-5D,5L Domain Scores
Description: General health status was assessed using the EQ-5D,5L questionnaire, which includes five dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 scoring levels, where 1 indicates a better health state (no problems) and 3 indicates a worse health state. A positive change indicates improvement.
Time Frame: EQ-5D,5L was assessed at baseline (Cycle 1 Day 1) and on Day 1 of every other cycle to Cycle 5 Day 1, every fourth cycle thereafter, beginning with Cycle 9 Day 1 and End of Treatment (EOT), up to 36 months. Each cycle is 21 days.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tebentafusp | Investigator's Choice
Number analyzed (Participants) | 252 | 126
Units on a scale
  Mobility - Baseline Cycle 1: number analyzed (Participants) | 194 | 78
  Mobility - Baseline Cycle 1 | 1.2 (0.62) | 1.3 (0.55)
  Mobility - Change at Cycle 3: number analyzed (Participants) | 136 | 45
  Mobility - Change at Cycle 3 | -0.1 (0.66) | 0.1 (0.47)
  Mobility - Change at Cycle 5: number analyzed (Participants) | 108 | 28
  Mobility - Change at Cycle 5 | 0.0 (0.73) | 0.3 (0.65)
  Mobility - Change at Cycle 9: number analyzed (Participants) | 71 | 14
  Mobility - Change at Cycle 9 | 0.0 (0.91) | 0.0 (0.55)
  Mobility - Change at Cycle 13: number analyzed (Participants) | 47 | 9
  Mobility - Change at Cycle 13 | -0.1 (0.60) | 0.3 (0.87)
  Mobility - Change at Cycle 17: number analyzed (Participants) | 22 | 6
  Mobility - Change at Cycle 17 | 0.3 (0.57) | 0.2 (0.41)
  Mobility - Change at Cycle 21: number analyzed (Participants) | 13 | 2
  Mobility - Change at Cycle 21 | 0.0 (0.58) | 0.5 (0.71)
  Mobility - Change at Cycle 25: number analyzed (Participants) | 8 | 1
  Mobility - Change at Cycle 25 | 0.1 (0.64) | 0.0 (0.00)
  Mobility - Change at Cycle 29: number analyzed (Participants) | 9 | 2
  Mobility - Change at Cycle 29 | 0.0 (0.50) | 0.0 (0.00)
  Mobility - Change at EOT: number analyzed (Participants) | 95 | 45
  Mobility - Change at EOT | 0.3 (0.73) | 0.4 (0.99)
  Self-care - Baseline Cycle 1: number analyzed (Participants) | 194 | 78
  Self-care - Baseline Cycle 1 | 1.1 (0.45) | 1.1 (0.29)
  Self-care - Change at Cycle 3: number analyzed (Participants) | 136 | 45
  Self-care - Change at Cycle 3 | 0.0 (0.49) | 0.0 (0.26)
  Self-care - Change at Cycle 5: number analyzed (Participants) | 108 | 28
  Self-care - Change at Cycle 5 | 0.0 (0.42) | 0.0 (0.00)
  Self-care - Change at Cycle 9: number analyzed (Participants) | 71 | 14
  Self-care - Change at Cycle 9 | 0.0 (0.58) | 0.0 (0.00)
  Self-care - Change at Cycle 13: number analyzed (Participants) | 47 | 9
  Self-care - Change at Cycle 13 | 0.1 (0.52) | 0.1 (0.33)
  Self-care - Change at Cycle 17: number analyzed (Participants) | 22 | 6
  Self-care - Change at Cycle 17 | 0.1 (0.68) | 0.0 (0.00)
  Self-care - Change at Cycle 21: number analyzed (Participants) | 13 | 2
  Self-care - Change at Cycle 21 | 0.0 (0.00) | 0.0 (0.00)
  Self-care - Change at Cycle 25: number analyzed (Participants) | 8 | 1
  Self-care - Change at Cycle 25 | 0.0 (0.00) | 0.0 (0.00)
  Self-care - Change at Cycle 29: number analyzed (Participants) | 9 | 2
  Self-care - Change at Cycle 29 | 0.0 (0.00) | 0.0 (0.00)
  Self-care - Change at EOT: number analyzed (Participants) | 95 | 45
  Self-care - Change at EOT | 0.1 (0.60) | 0.1 (0.56)
  Usual activities - Baseline Cycle 1: number analyzed (Participants) | 194 | 78
  Usual activities - Baseline Cycle 1 | 1.2 (0.53) | 1.3 (0.55)
  Usual activities - Change at Cycle 3: number analyzed (Participants) | 136 | 45
  Usual activities - Change at Cycle 3 | 0.2 (0.59) | 0.1 (0.73)
  Usual activities - Change at Cycle 5: number analyzed (Participants) | 108 | 28
  Usual activities - Change at Cycle 5 | 0.1 (0.61) | 0.2 (0.61)
  Usual activities - Change at Cycle 9: number analyzed (Participants) | 71 | 14
  Usual activities - Change at Cycle 9 | 0.2 (0.87) | 0.1 (0.53)
  Usual activities - Change at Cycle 13: number analyzed (Participants) | 47 | 9
  Usual activities - Change at Cycle 13 | 0.3 (0.79) | 0.1 (0.60)
  Usual activities - Change at Cycle 17: number analyzed (Participants) | 22 | 6
  Usual activities - Change at Cycle 17 | 0.5 (0.80) | 0.2 (0.41)
  Usual activities - Change at Cycle 21: number analyzed (Participants) | 13 | 2
  Usual activities - Change at Cycle 21 | 0.3 (0.48) | 0.0 (0.00)
  Usual activities - Change at Cycle 25: number analyzed (Participants) | 8 | 1
  Usual activities - Change at Cycle 25 | 0.3 (0.46) | 0.0 (0.00)
  Usual activities - Change at Cycle 29: number analyzed (Participants) | 9 | 2
  Usual activities - Change at Cycle 29 | 0.2 (0.44) | 0.0 (0.00)
  Usual activities - Change at EOT: number analyzed (Participants) | 95 | 45
  Usual activities - Change at EOT | 0.4 (0.77) | 0.5 (0.87)
  Pain/Discomfort - Baseline Cycle 1: number analyzed (Participants) | 194 | 78
  Pain/Discomfort - Baseline Cycle 1 | 1.5 (0.71) | 1.5 (0.73)
  Pain/Discomfort - Change at Cycle 3: number analyzed (Participants) | 136 | 45
  Pain/Discomfort - Change at Cycle 3 | 0.0 (0.75) | 0.1 (0.73)
  Pain/Discomfort - Change at Cycle 5: number analyzed (Participants) | 108 | 28
  Pain/Discomfort - Change at Cycle 5 | 0.0 (0.65) | 0.2 (0.72)
  Pain/Discomfort - Change at Cycle 9: number analyzed (Participants) | 71 | 14
  Pain/Discomfort - Change at Cycle 9 | 0.1 (0.73) | -0.1 (0.73)
  Pain/Discomfort - Change at Cycle 13: number analyzed (Participants) | 47 | 9
  Pain/Discomfort - Change at Cycle 13 | 0.1 (0.51) | 0.1 (0.93)
  Pain/Discomfort - Change at Cycle 17: number analyzed (Participants) | 22 | 6
  Pain/Discomfort - Change at Cycle 17 | 0.4 (0.85) | 0.3 (0.52)
  Pain/Discomfort - Change at Cycle 21: number analyzed (Participants) | 13 | 2
  Pain/Discomfort - Change at Cycle 21 | 0.2 (0.55) | 0.0 (0.00)
  Pain/Discomfort - Change at Cycle 25: number analyzed (Participants) | 8 | 1
  Pain/Discomfort - Change at Cycle 25 | 0.0 (0.53) | 1.0 (NA) — Not calculable due to single participant.
  Pain/Discomfort - Change at Cycle 29: number analyzed (Participants) | 9 | 2
  Pain/Discomfort - Change at Cycle 29 | 0.1 (0.60) | 0.5 (0.71)
  Pain/Discomfort - Change at EOT: number analyzed (Participants) | 95 | 45
  Pain/Discomfort - Change at EOT | 0.2 (0.87) | 0.4 (1.10)
  Anxiety/Depression - Baseline Cycle 1: number analyzed (Participants) | 194 | 78
  Anxiety/Depression - Baseline Cycle 1 | 1.8 (0.94) | 1.7 (0.89)
  Anxiety/Depression - Change at Cycle 3: number analyzed (Participants) | 136 | 45
  Anxiety/Depression - Change at Cycle 3 | -0.2 (0.77) | -0.3 (0.55)
  Anxiety/Depression - Change at Cycle 5: number analyzed (Participants) | 108 | 28
  Anxiety/Depression - Change at Cycle 5 | -0.2 (0.74) | 0.0 (0.61)
  Anxiety/Depression - Change at Cycle 9: number analyzed (Participants) | 71 | 14
  Anxiety/Depression - Change at Cycle 9 | -0.3 (0.80) | 0.1 (0.77)
  Anxiety/Depression - Change at Cycle 13: number analyzed (Participants) | 47 | 9
  Anxiety/Depression - Change at Cycle 13 | -0.4 (0.77) | -0.1 (0.60)
  Anxiety/Depression - Change at Cycle 17: number analyzed (Participants) | 22 | 6
  Anxiety/Depression - Change at Cycle 17 | -0.4 (0.85) | 0.0 (0.00)
  Anxiety/Depression - Change at Cycle 21: number analyzed (Participants) | 13 | 2
  Anxiety/Depression - Change at Cycle 21 | -0.5 (0.88) | 0.0 (0.00)
  Anxiety/Depression - Change at Cycle 25: number analyzed (Participants) | 8 | 1
  Anxiety/Depression - Change at Cycle 25 | -0.4 (0.74) | 0.0 (NA) — Not calculable due to single participant.
  Anxiety/Depression - Change at Cycle 29: number analyzed (Participants) | 9 | 2
  Anxiety/Depression - Change at Cycle 29 | -0.6 (0.88) | 0.5 (0.71)
  Anxiety/Depression - Change at EOT: number analyzed (Participants) | 95 | 45
  Anxiety/Depression - Change at EOT | 0.3 (0.94) | 0.2 (1.07)

5. Secondary Outcome: Quality-of-life: Change From Baseline in EQ-5D Visual Analogue Score (VAS)
Description: The EQ-5D VAS score records the participant's self-rated health on a vertical visual analogue scale, with 0 being the worst imaginable health state and 100 being the best imaginable health state. A positive change indicates improvement.
Time Frame: EQ-5D,5L VAS was assessed at baseline (Cycle 1 Day 1) and on Day 1 of every other cycle to Cycle 5 Day 1, every fourth cycle thereafter, beginning with Cycle 9 Day 1 and End of Treatment (EOT), up to 36 months. Each cycle is 21 days.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tebentafusp | Investigator's Choice
Number analyzed (Participants) | 252 | 126
Units on a scale
  Baseline Cycle 1: number analyzed (Participants) | 194 | 78
  Baseline Cycle 1 | 81.0 (16.36) | 80.4 (18.31)
  Change at Cycle 3: number analyzed (Participants) | 136 | 45
  Change at Cycle 3 | 0.4 (14.69) | -0.8 (14.28)
  Change at Cycle 5: number analyzed (Participants) | 108 | 28
  Change at Cycle 5 | 0.6 (15.61) | -0.7 (14.38)
  Change at Cycle 9: number analyzed (Participants) | 71 | 14
  Change at Cycle 9 | -0.9 (19.81) | -3.3 (13.30)
  Change at Cycle 13: number analyzed (Participants) | 47 | 9
  Change at Cycle 13 | -2.0 (16.48) | -2.6 (8.37)
  Change at Cycle 17: number analyzed (Participants) | 22 | 6
  Change at Cycle 17 | -10.2 (20.93) | -8.5 (33.82)
  Change at Cycle 21: number analyzed (Participants) | 13 | 2
  Change at Cycle 21 | -1.8 (14.52) | -1.0 (5.66)
  Change at Cycle 25: number analyzed (Participants) | 8 | 1
  Change at Cycle 25 | -13.6 (19.43) | -4.0 (NA) — Not calculable due to single participant
  Change at Cycle 29: number analyzed (Participants) | 9 | 2
  Change at Cycle 29 | 0.0 (9.25) | -2.0 (1.41)
  Change at EOT: number analyzed (Participants) | 95 | 45
  Change at EOT | -10.1 (22.53) | -11.7 (21.40)

6. Secondary Outcome: Quality-of-Life: Change From Baseline in EORTC QLQ-C30 Global Health Status
Description: Global health status and quality of life was assessed using the EORTC QLQ-C30 questionnaire. The score range for the EORTC QLQ-C30 is from 0 to 100, with higher scores indicating better functioning and better global health status and health-related quality of life. A positive change indicates improvement.
Time Frame: EORTC QLQ-C30 was assessed at baseline (Cycle 1 Day 1) and on Day 1 of every other cycle to Cycle 5 Day 1, every fourth cycle thereafter, beginning with Cycle 9 Day 1 and End of Treatment (EOT), up to 36 months. Each cycle is 21 days.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tebentafusp | Investigator's Choice
Number analyzed (Participants) | 252 | 126
Units on a scale
  Baseline Cycle 1: number analyzed (Participants) | 173 | 65
  Baseline Cycle 1 | 76.108 (20.233) | 74.872 (20.439)
  Change at Cycle 3: number analyzed (Participants) | 105 | 35
  Change at Cycle 3 | 0.952 (16.274) | -0.238 (14.919)
  Change at Cycle 5: number analyzed (Participants) | 94 | 22
  Change at Cycle 5 | -1.152 (20.797) | -10.227 (22.557)
  Change at Cycle 9: number analyzed (Participants) | 57 | 13
  Change at Cycle 9 | -2.193 (19.577) | -8.333 (13.176)
  Change at Cycle 13: number analyzed (Participants) | 40 | 9
  Change at Cycle 13 | -5.625 (17.641) | -10.185 (16.017)
  Change at Cycle 17: number analyzed (Participants) | 18 | 6
  Change at Cycle 17 | -10.185 (28.087) | -4.167 (6.972)
  Change at Cycle 21: number analyzed (Participants) | 11 | 2
  Change at Cycle 21 | 0.758 (18.429) | -4.167 (5.893)
  Change at Cycle 25: number analyzed (Participants) | 7 | 1
  Change at Cycle 25 | -2.381 (27.936) | 0.00 (0.00)
  Change at Cycle 29: number analyzed (Participants) | 6 | 1
  Change at Cycle 29 | -8.333 (19.720) | 0.00 (0.00)
  Change at EOT: number analyzed (Participants) | 76 | 34
  Change at EOT | -10.417 (20.911) | -10.539 (23.148)

7. Secondary Outcome: Pharmacokinetics (PK): Tebentafusp Concentration
Description: Serum PK concentrations of tebentafusp were collected over time.
Time Frame: PK concentrations were assessed at pre-dose, end of infusion and anytime in the 12 to 24 hour window after completion of the infusion in Cycle 1 on Days 1, 8 and 15.
Population: The PK Analysis Set included participants in the Safety Analysis Set who had at least 1 measurable PK concentration and who had relevant date, time, and dosing data for the sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tebentafusp
Number analyzed (Participants) | 231
pg/mL
  Cycle 1 Day 1 - End of Infusion: number analyzed (Participants) | 207
  Cycle 1 Day 1 - End of Infusion | 4201.929 (0.6)
  Cycle 1 Day 1 - 12 to 24 hours post-infusion: number analyzed (Participants) | 212
  Cycle 1 Day 1 - 12 to 24 hours post-infusion | 505.100 (0.7)
  Cycle 1 Day 8 - End of Infusion: number analyzed (Participants) | 200
  Cycle 1 Day 8 - End of Infusion | 5787.139 (0.4)
  Cycle 1 Day 8 - 12 to 24 hours post-infusion: number analyzed (Participants) | 198
  Cycle 1 Day 8 - 12 to 24 hours post-infusion | 738.602 (0.7)
  Cycle 1 Day 15 - End of Infusion: number analyzed (Participants) | 202
  Cycle 1 Day 15 - End of Infusion | 13715.914 (0.5)
  Cycle 1 Day 15 - 12 to 24 hours post-infusion: number analyzed (Participants) | 205
  Cycle 1 Day 15 - 12 to 24 hours post-infusion | 1685.354 (0.6)

8. Secondary Outcome: Efficacy: Objective Response Rate (ORR)
Description: Objective response rate (ORR) is defined as the proportion of patients achieving an objective response (RECIST v1.1).
Time Frame: ORR will be assessed after every participant has had at least 3 assessments, conducted every 3 months, up to 5.5 years.
Reporting Status: Not Posted

9. Secondary Outcome: Efficacy: Duration of Response (DOR)
Description: Duration of response (DOR) is defined as the time from first documented objective response (RECIST v1.1) until the date of documented disease progression.
Time Frame: DOR will be assessed every 3 months from randomization until disease progression, assessed up to 5.5 years.
Reporting Status: Not Posted

10. Secondary Outcome: Efficacy: Disease Control Rate (DCR)
Description: Disease control rate (DCR) is defined as the proportion of patients with either an objective response or stable disease (RECIST v1.1)
Time Frame: DCR will be assessed every 3 months from randomization until disease progression, up to 5.5 years.
Reporting Status: Not Posted

11. Secondary Outcome: Pharmacokinetics: Frequency of Anti-IMCgp100 Antibody Formation
Time Frame: Approximately 5 assessments will be performed between first dose of IMCgp100 and end of treatment, assessed up to 5.5 years.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 36 months.
Description: The Safety Analysis Set included all randomized participants who received at least 1 full or partial dose of tebentafusp or investigator's choice. Combining participants into a single group (Investigator's Choice) was pre-specified as part of the study design and data for each treatment in that arm were not analyzed separately. Adverse events were defined as events that were new or worsened during the on-treatment period.
Arm/Group | Tebentafusp | Investigator's Choice
All-Cause Mortality (participants affected / at risk) | 84/245 | 57/111
Serious Adverse Events (participants affected / at risk) | 69/245 | 26/111
Other Adverse Events (participants affected / at risk) | 245/245 | 102/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tebentafusp (N=245) | Investigator's Choice (N=111)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Hypopituitarism (Endocrine disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Periorbital edema (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (4) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (3) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 2 (2)
Biliary obstruction (Hepatobiliary disorders) | 1 (3) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 2 (18) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (3) | 3 (5)
Hypertransaminasemia (Hepatobiliary disorders) | 1 (5) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 24 (51) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Salmonella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Brain edema (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial mass (Nervous system disorders) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (2) | 0 (0)
Presyncope (Nervous system disorders) | 1 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Scrotal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (10) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (13) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 5 (6) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tebentafusp (N=245) | Investigator's Choice (N=111)
Anemia (Blood and lymphatic system disorders) | 25 (62) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 24 (51) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 6 (10)
Tachycardia (Cardiac disorders) | 24 (45) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 13 (16)
Hypothyroidism (Endocrine disorders) | 3 (3) | 12 (15)
Periorbital edema (Eye disorders) | 26 (51) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 59 (92) | 14 (21)
Abdominal pain upper (Gastrointestinal disorders) | 50 (79) | 14 (21)
Constipation (Gastrointestinal disorders) | 44 (65) | 13 (15)
Diarrhea (Gastrointestinal disorders) | 61 (120) | 22 (45)
Dry mouth (Gastrointestinal disorders) | 8 (9) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 20 (28) | 5 (5)
Nausea (Gastrointestinal disorders) | 119 (288) | 28 (44)
Vomiting (Gastrointestinal disorders) | 73 (163) | 10 (19)
Asthenia (General disorders) | 38 (71) | 9 (11)
Chills (General disorders) | 117 (378) | 4 (4)
Face edema (General disorders) | 25 (39) | 2 (2)
Fatigue (General disorders) | 124 (352) | 39 (53)
Influenza like illness (General disorders) | 18 (75) | 2 (2)
Edema peripheral (General disorders) | 66 (119) | 3 (3)
Pyrexia (General disorders) | 186 (682) | 7 (11)
Hepatic pain (Hepatobiliary disorders) | 15 (41) | 4 (4)
Hyperbilirubinemia (Hepatobiliary disorders) | 26 (56) | 6 (6)
Cytokine release syndrome (Immune system disorders) | 34 (91) | 0 (0)
Nasopharyngitis (Infections and infestations) | 20 (24) | 1 (1)
Urinary tract infection (Infections and infestations) | 14 (19) | 5 (5)
Alanine aminotransferase increased (Investigations) | 50 (127) | 12 (19)
Aspartate aminotransferase increased (Investigations) | 55 (134) | 11 (19)
Blood alkaline phosphatase increased (Investigations) | 23 (60) | 3 (4)
Blood creatinine increased (Investigations) | 13 (26) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 13 (20) | 3 (8)
Lipase increased (Investigations) | 35 (73) | 7 (12)
Weight decreased (Investigations) | 16 (16) | 7 (11)
Decreased appetite (Metabolism and nutrition disorders) | 45 (56) | 15 (17)
Hypokalemia (Metabolism and nutrition disorders) | 18 (24) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 19 (31) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 27 (52) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 53 (97) | 18 (30)
Back pain (Musculoskeletal and connective tissue disorders) | 45 (56) | 9 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 (30) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 24 (40) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (36) | 3 (3)
Dizziness (Nervous system disorders) | 26 (46) | 9 (12)
Headache (Nervous system disorders) | 75 (135) | 11 (15)
Parasthesia (Nervous system disorders) | 27 (53) | 1 (1)
Anxiety (Psychiatric disorders) | 13 (14) | 2 (2)
Insomnia (Psychiatric disorders) | 22 (24) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 44 (67) | 11 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 31 (42) | 7 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (22) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 77 (106) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 60 (120) | 1 (1)
Hair color changes (Skin and subcutaneous tissue disorders) | 48 (62) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 13 (17) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 168 (536) | 26 (33)
Rash (Skin and subcutaneous tissue disorders) | 132 (603) | 18 (25)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 75 (343) | 9 (10)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 51 (80) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 19 (24) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 22 (26) | 2 (2)
Vitiligo (Skin and subcutaneous tissue disorders) | 40 (45) | 4 (5)
Flushing (Vascular disorders) | 25 (34) | 1 (2)
Hypertension (Vascular disorders) | 38 (91) | 8 (8)
Hypotension (Vascular disorders) | 91 (212) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT03070392/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT03070392/SAP_001.pdf